CLINICAL TRIAL: NCT06844396
Title: The Impact of NICU Music Therapy on Preterm Infants' Clinical Markers and Caregiver Wellbeing
Brief Title: The Impact of NICU Music Therapy for Preterm Infants and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Collaborators: The Whittington Hospital NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ETH2425-0374
Record Dates: First submitted 2025-01-16; First posted 2025-02-25 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-10

CONDITIONS: Premature Birth
Keywords: NICU; Parent Mental Health; Music Therapy; Neonatal
MeSH Terms: conditions — Premature Birth | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music Therapy (Experimental): Music Therapy delivered twice weekly to infants on a NICU ward
  Interventions: Other: Music Therapy

INTERVENTIONS:
Other: Music Therapy — Music Therapy consisting of four types of protocol:
  * Music combined with skin to skin
  * Developmental multimodal technique
  * Infant directed singing
  * Parent/caregiver therapeutic support

SUMMARY:
This study aims to provide initial evidence for the use of music therapy in the NICU in a UK context. In other countries, such as the US and the Netherlands, music therapy is routinely provided in the NICU and research has demonstrated benefits for the both the child and their caregivers. As there is no existing UK-based research on music therapy in the NICU, medical institutions are reluctant to consider the benefits of music therapy. This reduces infants' access to non-invasive treatment in the NICU. Our study aims to address this gap.

DETAILED DESCRIPTION:
The aim of this pilot study is to investigate the impact of Neonatal Intensive Care Unit (NICU) Music Therapy (MT) interventions on preterm infants' clinical markers and caregiver wellbeing. The study will investigate changes in the participating infants' clinical markers (heart rate, oxygen saturation, blood pressure, respiration rate) before, during and after therapy, weight gain, feeding behaviours, sleep patterns, discharge time and caregiver wellbeing, including bonding and mood. The study also aims to assess the acceptability of music therapy for pre-term infants, caregivers and NICU staff, and explore how music therapy can be used on NICU wards in the UK.

NICU care, while lifesaving, has been shown to have negative long-term consequences, which can include repeated activation of the stress response and reduced maternal interaction, with possible negative long-term impacts on brain development.

The NHS published an action plan to implement recommendations for improving neonatal care. The report does not specify music therapy. However, initial research in the US, Switzerland, and the Netherlands has shown clinically and statistically significant improvements on well-being, stress reduction and neural development in the neonate. Beyond these crucial findings, music therapy had a positive effect on parent well-being, parent-child interaction and the overall reduction of noise levels on the ward.

This pilot study will consist of a six-week data collection period. During this time, infants and their primary caregiver(s) will be invited to participate in the study on admission to the NICU.

Participants will be offered music therapy sessions twice weekly over the course of the six-week data collection period. The music therapist will determine the appropriate music therapy interventions according to the infant's needs, therapeutic goals and corrected gestational age. These could include one of the four interventions from the NICU-MT method depending on therapeutic need, 1) music combined with caregiver skin to skin, 2) developmental multimodal technique, 3) infant directed singing and 4) caregiver therapeutic support. The caregiver may also be involved in the session during the use of multimodal technique, infant directed singing, and caregiver skin to skin. Sessions will last approximately 30 minutes, with 10 - 20 minutes of music.

NICU staff working on the ward during the study and caregivers will also be invited to participate in the evaluation of the acceptability of the music therapy intervention.

The quantitative data from infants participating in this study will comprise of routine data gathered for clinical purposes. The investigators will use data gathered at the time of the music therapy intervention and during a control time (no intervention) to measure the impact of the intervention on clinical markers. Data routinely collected at the High Dependency Unit (HDU) includes hourly recording on an observation sheet of temperature, heart rate, respiratory rate and oxygen saturations using Nellcor/Covidien monitors.

The study will also gather data relating to feeding behaviours, weight gain, length of stay and sleep patterns as well as follow up data relating to developmental milestones.

To assess bonding and emotional wellbeing, parents will be asked to complete three questionnaires before the first music therapy session and after the last music therapy session.

To investigate how music therapy is used with pre-term infants and their families in the NICU, the music therapist will keep a log of music therapy interventions used, including clinical notes relating to infant and family responses during the session. They will also complete a fidelity checklist after each session, for the purposes of monitoring adherence to the interventions outlined in the protocol.

Ultimately, this pilot study will inform and support further research in this area focusing on longer-term outcomes for NICU infants. As there is no UK-based evidence for the use of NICU-MT on wards in the UK, medical institutions are unwilling to consider the benefits of music therapy as standard for infant care. This sets the UK far behind other countries in terms of non-invasive treatments for this population.

ELIGIBILITY:
Infant Participants:

Inclusion Criteria:

* Infants in or admitted to the Whittington NHS Trust NICU High Dependency Unit (HDU) during the 6-week intervention and data collection period
* Infants are medically stable
* Infants at 28 weeks corrected gestational age and above

Exclusion Criteria:

* Infants who are medically unstable
* Infants younger than 28 weeks CGA
* Severe hearing impairment or hearing loss

Primary Caregivers:

Inclusion criteria:

* Primary caregiver(s) of an infant participating in the study
* Ability to complete questionnaires in English

NICU Staff

Inclusion criteria:

* 1 month experience working at the Whittington NHS Trust NICU
* At least two days' experience working on music therapy service provision days during the intervention period

Min Age: 28 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Infant Temperature | Baseline (resting state), within 15 minutes pre-intervention, during the intervention, within 15 minutes post-intervention, and periprocedurally
  Routinely collected clinical data will be collected for each infant participant to include temperature reported at degrees celcius. The data is collected using Nellcor/Covidien monitors
Infant Heart Rate | Baseline (resting state), within 15 minutes pre-intervention, during the intervention, within 15 minutes post-intervention, and periprocedurally
  Routinely collected clinical data will be collected for each infant participant to include heart rate reported in beats per minute. The data is collected using Nellcor/Covidien monitors
Infant Respiratory Rate | Baseline (resting state), within 15 minutes pre-intervention, during the intervention, within 15 minutes post-intervention, and periprocedurally
  Routinely collected clinical data will be collected for each infant participant to include respiratory rate reported in breaths per minute. The data is collected using Nellcor/Covidien monitors
Infant Oxygen Saturation | Baseline (resting state), within 15 minutes pre-intervention, during the intervention, within 15 minutes post-intervention, and periprocedurally
  Routinely collected clinical data will be collected for each infant participant to include oxygen saturation reported by percentage. The data is collected using Nellcor/Covidien monitors

SECONDARY OUTCOMES:
Infant Calorie Intake | Weeks 1 - 6 of the study period, or as long as the infant is admitted to NICU during the 6 week period.
  • Data relating to feeding behaviours will be recorded in caloric intake and reported in ml daily throughout the intervention period.
Infant Weight | Weeks 1 - 6 of the study period, or as long as the infant is admitted to NICU during the 6 week period.
  Data relating to weight gain in kg will be recorded daily throughout the intervention period
Infant Sleep Record | Weeks 1 - 6 of the study period, or as long as the infant is admitted to NICU during the 6 week period.
  • Data relating to sleeping patterns will be recorded in hours and reported daily throughout the intervention period.
Infant Length of Hospital Stay | From enrollment to the end of the infant's treatment or at 6 weeks
  • Data relating to length of hospital stay will be recorded in days.
Caregiver Postpartum Bonding Questionnaire | Weeks 1 - 6 of the study period, or as long as the infant is admitted to NICU during the 6 week period.
  • To assess bonding and emotional wellbeing, parents will be asked to complete the Postpartum Bonding Questionnaire (PBQ) immediately before the first intervention and immediately after the last intervention. The PBQ has 25 statements, each followed by six alternative responses ranging from 'always' to 'never'. Positive responses, such as ''I enjoy playing with my baby'', are scored from zero ('always') to 5 ('never'). Negative responses, such as ''I am afraid of my baby'', are scored from 5 ('always') to zero ('never'). The scores are summated for each factor, a high score indicating pathology.
Caregiver Perceived Stress Scale-NICU | Weeks 1 - 6 of the study period, or as long as the infant is admitted to NICU during the 6 week period.
  • To assess bonding and emotional wellbeing, parents will be asked to complete the Perceived Stress Scale-NICU (PSS-NICU) immediately before the first intervention and immediately after the last intervention. The PSS-NICU asks the parent to rate a variety of sights and sounds, their baby's looks and behaviour, their parental role and relationship with the baby, and staff behaviour and communication on a scale of N/A, not at all stressful, a little stressful, moderately stressful, very stressful and extremely stressful. The higher the score, the more stressed a parent is feeling.
Caregiver State-Trait Anxiety Inventory | Weeks 1 - 6 of the study period, or as long as the infant is admitted to NICU during the 6 week period.
  • To assess bonding and emotional wellbeing, parents will be asked to complete the State-Trait Anxiety Inventory (STAI-6) immediately before the first intervention and immediately after the last intervention. The questionnaire asks respondents to select the most appropriate response to 20 statements relating to anxiety: 1 (not at all) 2 (a little) 3 (somewhat) or 4 (very much so). Some questions are reverse coded and therefore some questions indicate anxiety if they are given a high score, whereas reverse coded questions indicate anxiety if they are given a low score.

OTHER OUTCOMES:
Acceptability of NICU Music Therapy | Weeks 1 - 6 of the study period, or as long as the infant is admitted to NICU during the 6 week period.
  Participating caregivers and NICU staff will be invited to complete a questionnaire about their experiences with music therapy on the NICU. The questionnaire comprises of statements and open questions to gather quantitative and qualitative information. The questions are as follows:
  What do you think about having music therapy on the ward? (options given) To what extent did music therapy affect infant responses? (options given) How would you rate your responses to music therapy on the ward? (options given) What benefits do you think could result from having music therapy on the ward? (open question) What challenges do you think could result from having music therapy on the ward? (open question) Would you recommend music therapy to other parents or carers on the ward during their stay? (options given)
Music Therapy Intervention Fidelity | Weeks 1 - 6 of the study period.
  The music therapist will utilise a fidelity checklist to monitor which music interventions were used and the extent to which the music therapy sessions adhered to or deviated from interventions outlined in the protocol, namely the four music therapy protocols drawn from the NICU-MT method. The fidelity checklist requires the therapist to record the following information for each music therapy session they provide for each infant participating in the study: Eligibility Checklist complete? (Y/N) Parent/ Carer Consent? (Y/N) MT Interventions Used (i.e. skin to skin, multimodal, singing, parent therapeutic support Resources and Equipment Length of session Time/Date Caregiver/s involved? Y/N Infant Responses (i.e. regulation, tolerance, sleep) Caregiver Responses (i.e. Mood, wellbeing state or caregiver/infant interaction Other Notes (deviations from protocol, interruptions or medical interventions at the same time, explaining changes in infant and why?)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Pool, PhD, Principal Investigator — Anglia Ruskin University
Locations (1):
- Whittington NHS Health Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside of the sponsor organisation and will be kept securely within internal University secure sharing systems.

REFERENCES:
- [Background] Walworth D, Standley J, Robertson A, Smith A, Swedberg O, Peyton JJ. (2012). Effects of neurodevelopmental stimulation on premature infants in neonatal intensive care: Randomized controlled trial. Journal of Neonatal Nursing, 18, 210-216.
- [Background] Whipple, J. (2005). Music and multimodal stimulation as developmental interven- tion in neonatal intensive care. Music Therapy Perspectives, 23(2), 100-105.
- [Background] Whipple J. The effect of parent training in music and multimodal stimulation on parent-neonate interactions in the neonatal intensive care unit. J Music Ther. 2000 Winter;37(4):250-68. doi: 10.1093/jmt/37.4.250. PMID 11281808
- [Background] Standley J. Music therapy research in the NICU: an updated meta-analysis. Neonatal Netw. 2012 Sep-Oct;31(5):311-6. doi: 10.1891/0730-0832.31.5.311. PMID 22908052
- [Background] Standley JM, Cassidy J, Grant R, Cevasco A, Szuch C, Nguyen J, Walworth D, Procelli D, Jarred J, Adams K. The effect of music reinforcement for non-nutritive sucking on nipple feeding of premature infants. Pediatr Nurs. 2010 May-Jun;36(3):138-45. PMID 20687305
- [Background] Standley JM. The effect of music and multimodal stimulation on responses of premature infants in neonatal intensive care. Pediatr Nurs. 1998 Nov-Dec;24(6):532-8. PMID 10085995
- [Background] Standley, J.M. and Gutierrez, C., 2020. Benefits of a Comprehensive Evidence-Based NICU-MT Program: Family-Centered, Neurodevelopmental Music Therapy for Premature Infants. Pediatric Nursing, 46(1).
- [Background] Miles MS, Funk SG, Carlson J. Parental Stressor Scale: neonatal intensive care unit. Nurs Res. 1993 May-Jun;42(3):148-52. PMID 8506163
- [Background] Marteau TM, Bekker H. The development of a six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI). Br J Clin Psychol. 1992 Sep;31(3):301-6. doi: 10.1111/j.2044-8260.1992.tb00997.x. PMID 1393159
- [Background] Jaschke, A.C. (2020), Muziektherapeutisch interventies 3.0 - How to hack the academy?, Special Issue, Tijdschrift voor Vaktherapie 16(4)
- [Background] Ormston K, Howard R, Gallagher K, Mitra S, Jaschke A. The Role of Music Therapy with Infants with Perinatal Brain Injury. Brain Sci. 2022 Apr 29;12(5):578. doi: 10.3390/brainsci12050578. PMID 35624965
- [Background] Detmer, M.R. (2016b). The use of parental singing: Enhancing neurodevelopment in premature infants. Imagine, 7(1), 66- 69.
- [Background] Cevasco-Trotter AM, Hamm EL, Yang X, Parton J. Multimodal Neurological Enhancement Intervention for Self-regulation in Premature Infants. Adv Neonatal Care. 2019 Aug;19(4):E3-E11. doi: 10.1097/ANC.0000000000000595. PMID 30946037
- [Background] Cevasco AM. The effects of mothers' singing on full-term and preterm infants and maternal emotional responses. J Music Ther. 2008 Fall;45(3):273-306. doi: 10.1093/jmt/45.3.273. PMID 18959452
- [Background] Brockington IF, Fraser C, Wilson D. The Postpartum Bonding Questionnaire: a validation. Arch Womens Ment Health. 2006 Sep;9(5):233-42. doi: 10.1007/s00737-006-0132-1. Epub 2006 May 4. PMID 16673041
- [Background] van Dokkum, N.H., Kooi. E.M.W., Berhane, B., Ravensbergen, A.G., Hakvoort, L., Jaschke, A.C. & Bos, A.F., (2021), Neonatal music therapy and cerebral oxygenation in extremely and very preterm infants: a pilot study, Special Issue 13(2): Music Therapy in the Neonatal Intensive Care Unit
- [Background] van Dokkum NH, Jaschke AC, Ravensbergen AG, Reijneveld SA, Hakvoort L, de Kroon MLA, Bos AF. Feasibility of Live-Performed Music Therapy for Extremely and Very Preterm Infants in a Tertiary NICU. Front Pediatr. 2020 Oct 16;8:581372. doi: 10.3389/fped.2020.581372. eCollection 2020. PMID 33178653
- [Background] Anderson DE, Patel AD. Infants born preterm, stress, and neurodevelopment in the neonatal intensive care unit: might music have an impact? Dev Med Child Neurol. 2018 Mar;60(3):256-266. doi: 10.1111/dmcn.13663. Epub 2018 Jan 24. PMID 29363098
- [Background] Span LC, van Dokkum NH, Ravensbergen AG, Bos AF, Jaschke AC. Combining Kangaroo Care and Live-Performed Music Therapy: Effects on Physiological Stability and Neurological Functioning in Extremely and Very Preterm Infants. Int J Environ Res Public Health. 2021 Jun 18;18(12):6580. doi: 10.3390/ijerph18126580. PMID 34207310
- [Background] Kraft KE, Jaschke AC, Ravensbergen AG, Feenstra-Weelink A, van Goor MEL, de Kroon MLA, Reijneveld SA, Bos AF, van Dokkum NH. Maternal Anxiety, Infant Stress, and the Role of Live-Performed Music Therapy during NICU Stay in The Netherlands. Int J Environ Res Public Health. 2021 Jul 2;18(13):7077. doi: 10.3390/ijerph18137077. PMID 34281014
- [Background] Bos M, van Dokkum NH, Ravensbergen AG, Kraft KE, Bos AF, Jaschke AC. Pilot study finds that performing live music therapy in intensive care units may be beneficial for infants' neurodevelopment. Acta Paediatr. 2021 Aug;110(8):2350-2351. doi: 10.1111/apa.15867. Epub 2021 May 2. No abstract available. PMID 33811376